CLINICAL TRIAL: NCT07252271
Title: Very Low Dose, add-on Prednisolone in Patients With Newly Diagnosed Rheumatoid Arthritis: a Randomised Placebo-controlled Study
Brief Title: Very Low Dose Prednisolone on Newly Diagnosed Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho SO, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VlP
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Rhematoid Arthritis
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- very low dose prednisolone (Active Comparator): Randomization will be performed using a computer-generated randomization list provided by the research pharmacist, adopting a permuted blocks design with block sizes of 4. Allocation concealment will be ensured by the use of sequentially numbered, opaque, sealed envelopes. Treatment will be masked to patients and investigators. The participants will be instructed to take the study drugs daily for 10 weeks. For the prednisolone group, the dose of the active drug will be 4mg once daily for 4 weeks then tapering at 1mg/week every 2-week till off at week 10.
  Interventions: Drug: Prednisolone
- Control (Placebo Comparator): Randomization will be performed using a computer-generated randomization list provided by the research pharmacist, adopting a permuted blocks design with block sizes of 4. Allocation concealment will be ensured by the use of sequentially numbered, opaque, sealed envelopes. Treatment will be masked to patients and investigators. The participants will be instructed to take the study drugs daily for 10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — The dose prednisolone will be 4mg once daily for 4 weeks then tapering at 1mg/week every 2-week till off at week 10.
  Arms: very low dose prednisolone
Drug: Placebo — The dose of placebo will be 4mg once daily for 4 weeks then tapering at 1mg/week every 2-week till off at week 10.
  Arms: Control

SUMMARY:
Objective To investigate the efficacy of prednisolone 4mg/day added to standard of care in newly diagnosed rheumatoid arthritis (RA) patients with active disease.

Hypothesis Add-on prednisolone 4mg/day is efficacious compared to placebo in newly diagnosed RA patients with active disease.

Design and subjects This is a 12-week, randomized, placebo-controlled, double-blind study. We plan to enroll 112 adult patients with newly diagnosed active RA (Disease Activity Score 28-C-Reactive Protein [DAS28-CRP] > 3.2). They will be randomized 1:1 to receive prednisolone 4mg once daily for 5 weeks then tapering at 1mg/week each week till off or placebo. Conventional synthetic disease-modifying-anti-rheumatic-drugs (DMARDs) will be started and adjusted according to a standard protocol aiming to achieve low disease activity. Patients with contra-indications to prednisolone, or requiring biologic or targeted synthetic DMARDs will be excluded.

Study instruments Clinical response will be monitored using DAS28-CRP every 4 weeks. Adverse events (AE), severe AE (SAE) and AE of special interest (AESI) will be recorded at every visit.

Main outcome measures and analysis The primary outcome is the change of DAS28-CRP comparing the two groups at week-4 by student T test. Secondary outcomes include the changes of DAS28-CRP at week-8 and week-12 as well as proportion of patients with AE comparing the two groups. Independent factors predicting disease control will be analyzed by multivariate logistic regression.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of prednisolone 4mg/day added to standard of care in terms of disease activity control in newly diagnosed RA patients with active disease. It is hypothezed add-on prednisolone 4mg/day is efficacious compared to placebo in newly diagnosed RA patients with active disease in the short-term.

This is an investigator-initiated, single-center, randomized, placebo-controlled, double-blind study. The intervention duration is 10 weeks. The follow-up period is 24 weeks. The recruitment period is 30 months. The total study duration will be 3 years.

All the participants (n=112) will be randomized in a 1:1 ratio to prednisolone (n=56) or placebo (n=56) group. Randomization will be performed using a computer-generated randomization list provided by the research pharmacist, adopting a permuted blocks design with block sizes of 4.

Allocation concealment will be ensured by the use of sequentially numbered, opaque, sealed envelopes. Treatment will be masked to patients and investigators. The participants will be instructed to take one study capsule (prednisolone or placebo) daily for 10 weeks. For the prednisolone group, the dose of the active drug will be 4mg once daily for 4 weeks then tapering at 1mg/week every 2-week till off at week 10. All participants will also be given csDMARDs and treated to a target of DAS28 low disease activity (<3.2) at Prince of Wales Hospital (PWH) throughout the study period according to a standard protocol modified to our study based on the EULAR recommendation and the Hong Kong guideline on the use of DMARDs (Figure 2). Disease activity and adverse events will be monitored at 4 weeks, 8 weeks, 12 weeks and 24 weeks. Patients will be advised to reach out to the rheumatologists earlier if the condition changes unexpectedly. Changes in the dosage or addition of nonsteroidal antiinflammatory drugs are allowed. Switching to a new csDMARD is possible in case of toxicity or intolerance. The use of b/tsDMARDs or additional systemic GC will be prohibited throughout the study. All medication changes will be documented in detail. Participants who required rescue b/tsDMARDs or systemic GC will be withdrawn from the study. They will be treated according to the standard of care with regular assessment till the end of the study. All patients will be given calcium and vitamin D supplements throughout the study period. The following clinical variables will be assessed at each visit: erythrocyte sedimentation rate(ESR), CRP, number of swollen joints (0-28), number of tender joints (0-28), visual analogue scale (VAS) for pain (0-100 mm=most pain), VAS for patient's global assessment (0-100 mm=worst score), VAS for physician's global assessment (0-100 mm=worst score), and DAS28 score. The presence of rheumatoid factor (RF) and cyclic citrullinated peptide (CCP) antibody with their respective serum levels will be documented at baseline. The number of damaged joints will be assessed at baseline and the end of the study. Rheumatoid factor status and anti-cyclic citrullinated peptide antibodies status will be determined at baseline. Functional disability is assessed by the disability index of HAQ (0-3=most functional disability). ACR20/50/70 responses are defined as at least 20%, 50%, and 70% improvement in swollen joint and tender joint counts, and three of five other variables (i.e., ESR or CRP, HAQ score, pain score, and physicians' and patients' global assessments). All assessments and consultations will be done by rheumatologists (investigators) with more than 10 years experience. Preparation of study medications Both the active drug (prednisolone) and placebo will be repackaged into capsules with identical appearance according to the standard operating procedure of the Clinical Research Pharmacy, School of Pharmacy, The Chinese University of Hong Kong. On entering the trial, each participant will be given a filled and labeled bottle, coded with a unique study number, which will be used for all future supplies of study drugs for that patient. Study treatment will remain masked for the patients, investigators, and study personnel throughout the trial. Code breaking is allowed in special circumstances by informing the Clinical Research Pharmacy or at end of the study.

Toxicity monitoring To monitor the possible side effect of prednisolone and other medications, complete blood count, liver function test and renal function test will be performed at screening, week 4, week 8, week 12 and week 24. Body mass index, blood pressure, blood sugar and lipid profile will be checked at baseline, week 4, week 8, week 12 and week 24. Chest x-rays will be obtained at screening and when clinically indicated. Hepatitis status and electrocardiogram will be done at screening.

The treating physicians will record all adverse events (AEs) and, if necessary, make treatment adjustments in accordance with the protocol. Serious AEs (SAEs) are defined as the occurrence of life-threatening condition or death, a significant or permanent disability, a malignancy, hospitalization or prolongation of hospitalization, a congenital abnormality, or a birth defect. AEs of special interest (AESI) will also be collected which include any AE leading to drug discontinuation, MACE (myocardial infarction, cerebrovascular or peripheral arterial vascular event), newly occurring hypertension/diabetes/infection/cataract/glaucoma and fragility fracture.

Consecutive RA patients attending the rheumatology clinics of PWH, Tai Po Hospital (TPH), Alice Ho Miu Ling Nethersole Hospital (AHNH), Princess Margaret Hospital (PMH) and Pamela Youde Nethersole Eastern Hospital (PYNEH) will be screened for eligibility. The inclusion criteria are: 1) ≥18 year-old, 2) fulfilment of the 2010 ACR/EULAR classification criteria of RA, 3) never use of any DMARDs for RA, and 4) disease activity score 28-C-reactive protein (DAS28-CRP) >3.2. The exclusion criteria are: 1) pregnancy or premenopausal women planning pregnancy, 2) functional status class IV (limited in ability to perform usual self-care, vocational, and avocational activities), 3) use of systemic GC in recent one month, and 4) contraindications to prednisolone.

A total of 112 patients who meet the criteria will be included (figure 3). A sample size determination was conducted for the primary outcome measurement, the difference in the change of DAS28-CRP at 4 weeks comparing the 2 groups, using Power Analysis and Sample Size Software (PASS version 11). From the published results of the GLORIA trial, the short-term (3 months) improvement in DAS28 in the prednisolone group and placebo group was 1.36±1.14 (baseline 4.40±1.04) and 0.73±1.21 (baseline 4.46±0.99) respectively (21). In our pilot study mentioned above, the improvement in mean DAS28 was - 1.4 ± 1.3 post-treatment. Therefore, more conservatively, we expect the difference of the change of DAS28-CRP at 4 weeks to be 0.6 comparing the prednisolone and placebo group. At least 49 patients will be required in each group to achieve a statistical power of 0.8 with a two-sided α of 0.05. With an estimated dropout rate of 15%, a total sample size of 112 would be required.

The study will be submitted to The Joint Chinese University of Hong Kong - New Territories East Cluster Clinical Research Ethics Committee and the Central Institutional Research Board of the Hospital Authority for approval. It will also be submitted to the clinicaltrials.gov for registration.

Written informed consent will be obtained from all participants prior to any of the trial procedure.

The study will be conducted according to the Declaration of Helsinki and ICH-GCP guidelines.

(iv) Data processing and analysis Patients who discontinue treatment or violate treatment protocol will be excluded from the analysis (per-protocol analysis). Missing data are assumed missing at random and will be treated using a multiple imputation method. Descriptive statistics will be used to present the baseline demographic and clinical variables included frequencies, means with standard deviations and median with interquartile range. T-test or Mann-Whitney U test and Chi-square test or fisher exact test will be used to evaluate the differences in clinical variables between the prednisolone and the placebo group at baseline, depending on the data distribution. The primary outcome measurement, the difference in the change of DAS28-CRP at 4 weeks comparing the 2 groups, will be analyzed by T-test. Clinical variables which are significantly different between the 2 groups in the univariate analyses and are biologically plausible (eg. age, sex, disease duration, disease activity or treatment) will be adjusted in the multivariate regression model to confirm the prednisolone treatment effect. The secondary outcomes on disease activity at week 8, week 12 and week 24 or disability in terms of HAQ at different time points will be compared likewise. The within group changes of these measurements before and after treatment will be examined using paired t-test or Wilcoxon signed-rank test. To look for the changes across study period across 2 groups, the repeated ANOVA test will be performed. To address the secondary outcome ofcomparison of proportion of patients with AE in the 2 groups, Chi-square test will be performed and cross-checked by generalized estimating equation (GEE) analysis. Independent factors predicting treatment response in terms of achieving low disease activity or remission at week 4 will be analysed by multivariate logistic regression. Sensitivity analysis using an intention-to-treat approach including all randomized patients will be done. A 2-tailed probability value of p<0.05 is considered statistically significant. Calculation will be performed using IBM SPSS Statistics Version 24 (IBM, Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 year-old
2. Fulfilment of the 2010 ACR/EULAR classification criteria of RA
3. Never use of any DMARDs for RA -

Exclusion Criteria:

1. Pregnancy or premenopausal women planning pregnancy
2. Functional status class IV (limited in ability to perform usual self-care, vocational, and avocational activities)
3. Use of systemic GC in recent one month
4. Contraindications to prednisolone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
the change of DAS28-CRP at 4 weeks comparing prednisolone group and placebo group. | 4 weeks
  DAS28-CRP is a composite score of CRP, patient global VAS, tender joint count and swollen joint count

SECONDARY OUTCOMES:
Changes of RA disease activity (DAS28-CRP) at week-8, week-12 and week 24 comparing the 2 groups. | 24 weeks
  Disease activity will be monitored at Week 4, Week 8, Week 12, and Week 24.
Changes of RA disease activity (DAS28-CRP) at different time points within the 2 groups. | 24 weeks
  Disease activity will be monitored at Week 4, Week 8, Week 12, and Week 24.
Disability at different time points comparing the 2 groups. | 24 weeks
  Functional disability is assessed by the disability index of HAQ (0-3=most functional disability) at week 4, week 8, week 12 and week 24. Comparison will be made between prednisolone and placebo group.
  The disability in terms of HAQ at different time points comparing the 2 groups, will be analyzed by T-test.
Proportion of patients with adverse events comparing the 2 groups. | 24 weeks
  We will record all adverse events (AEs) and, if necessary, make treatment adjustments in accordance with the protocol. Serious AEs (SAEs) are defined as the occurrence of life-threatening condition or death, a significant or permanent disability, a malignancy, hospitalization or prolongation of hospitalization, a congenital abnormality, or a birth defect. AEs of special interest (AESI) will also be collected which include any AE leading to drug discontinuation, MACE (myocardial infarction, cerebrovascular or peripheral arterial vascular event), newly occurring hypertension/diabetes/infection/cataract/glaucoma and fragility fracture.
  To address the secondary outcome of comparison of proportion of patients with AE in the 2 groups, Chi-square test will be performed and cross-checked by generalized estimating equation (GEE) analysis.
Independent predictors of RA disease control in all participants | 24 weeks
  Independent clinical factors predicting treatment response in terms of achieving low disease activity or remission at week 4 will be analysed by multivariate logistic regression

DOCUMENTS (1):
  • Study Protocol (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT07252271/Prot_000.pdf